CLINICAL TRIAL: NCT06841055
Title: A Phase II, Multisite, Open-label, Single Arm Trial of BNT327 in Combination With Docetaxel in Second-line Stage IV Non-small Cell Lung Cancer (NSCLC) Following Chemoimmunotherapy
Brief Title: Safety and Preliminary Effectiveness of BNT327, an Investigational Therapy for Patients With Non-small Cell Lung Cancer in Combination With Chemotherapy Following Chemoimmunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-07; 2024-518279-80-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Second-line treatment; Immunotherapy; Combination with other investigational agents; Bispecific antibody; Vascular endothelial growth factor (VEGF) A; Programmed death-ligand 1 (PD-L1); Combination with chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A - Pumitamig Dose 1 + docetaxel (Experimental)
  Interventions: Drug: Pumitamig; Drug: Docetaxel
- Part 1B - Pumitamig Dose 2 + docetaxel (Experimental)
  Interventions: Drug: Pumitamig; Drug: Docetaxel
- Part 2 - Selected doses of pumitamig + docetaxel (Experimental): Dose expansion at the deemed safe dose
  Interventions: Drug: Pumitamig; Drug: Docetaxel

INTERVENTIONS:
Drug: Pumitamig — Intravenous infusion
  Other Names: BNT327
Drug: Docetaxel — Intravenous infusion

SUMMARY:
This is a Phase II, multisite, open-label, single arm study with two parts in participants with advanced/metastatic NSCLC which progressed after a first-line chemoimmunotherapy.

Part 1 is safety run-in with pumitamig (BNT327) (Dose 1 or Dose 2) plus docetaxel and will include up to 12 participants to be treated in Part 1A and 1B sequentially.

Part 2 is a dose expansion at the deemed safe dose of pumitamig plus docetaxel.

DETAILED DESCRIPTION:
If the dose level (either from Part 1A or 1B) seems tolerable, an internal review committee will decide if the study can proceed to Part 2 and enroll additional participants.

Study participants will receive pumitamig in combination with docetaxel until disease progression, the occurrence of intolerable toxicity, study participant withdrawal, death, study termination or 2-year limit (whichever comes first).

After completion of study treatment, except for participants who withdraw informed consent, a long-term follow-up will be conducted for all participants to record disease progression, subsequent new anticancer treatments, and survival status.

ELIGIBILITY:
Key Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of Stage IV NSCLC that has documented radiographic progression on one or after one prior line of systemic treatment (programmed death-1 [PD-1]/ programmed death ligand-1 [PD-L1] inhibitor and platinum-based chemotherapy concomitantly) in advanced/metastatic setting per the American Joint Committee on Cancer staging system, 8th edition.

  * Participants must have received minimum two cycles of immunotherapy in first-line treatment to be eligible to this trial.
  * Only one prior line of immunotherapy containing regimen is allowed in advanced/metastatic setting. If participant had received adjuvant immunotherapy the disease-free interval (after the last dose of adjuvant immunotherapy) should be at least 6 months.
  * Historical PD-L1 results must be available.
  * Patients with actionable genetic alterations are allowed to be enrolled if patients received locally approved and available targeted agent in combination with immunotherapy in first-line advanced/metastatic setting.
  * Enrollment of participants with primary resistance (best response being radiological progression to prior immunochemotherapy) will be capped under 30% in the overall trial population.
* Have at least one measurable lesion as the targeted lesion based on RECIST v1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been documented after irradiation. Historical images within 28 days of the Screening Visit may be accepted as a screening image if deemed acceptable in the opinion of the investigator.
* Eastern cooperative oncology group performance status of 0 or 1.
* Adequate organ function.

Key Exclusion Criteria:

* Known hypersensitivity to the study treatments, their metabolites or formulation of excipients including polysorbate 80 (see Docetaxel label).
* Participants who received prior treatment with anti-vascular endothelial growth factor (VEGF) monoclonal antibody, or anti-PD-(L)-1/aVEGF bispecific antibody or docetaxel as monotherapy or in combination with other agents.
* Have received more than one prior lines of therapies in advanced/metastatic setting.
* Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 14 days prior to the initiation of study treatment (except for docetaxel premedication). Note: local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens) are allowed.
* Have uncontrolled hypertension or poorly controlled diabetic conditions prior to study treatment.
* Have a serious non-healing wound, ulcer, or bone fracture. This includes history (within 6 months prior to study entry) or risk of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra abdominal abscess or esophageal and gastric varices, or acute gastrointestinal bleeding. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Participants with evidence of major coagulation disorders or other significant risks of hemorrhage.
* Have superior vena cava syndrome or symptoms of spinal cord compression

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Occurrence of DLTs | up to 21 days after first dose of investigational medicinal product (IMP)
  During the DLT evaluation period by dose level
Part 1 and Part 2 - Occurrence of pumitamig treatment emergent adverse events (TEAEs), treatment-related TEAEs, treatment emergent serious adverse events (TESAEs), treatment-related (TRSAEs), and adverse events of special interest (AESIs) | from initiation of the first dose of IMP to the 90-day Follow-Up visit
  Graded according to the (US) National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Part 1 and Part 2 - Occurrence of dose interruption, dose reduction, and/or participant discontinuation due to adverse events (AEs) | from initiation of the first dose of IMP until the 90-day Safety Follow-up visit
Part 1 and Part 2 - Objective response rate (ORR) | Up to approximately 2 years
  Defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) based on investigator's review) is observed as best overall response

SECONDARY OUTCOMES:
Part 1 and Part 2 - Duration of Response (DOR) | Up to approximately 2 years
  Defined as the time from first objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) to first occurrence of objective tumor progression (progressive disease, per RECIST v1.1 based on the investigator's assessment) or death from any cause, whichever occurs first
Part 1 and Part 2- Progression-free Survival (PFS) | Up to approximately 2 years
  Based on the investigator's assessment defined as the time from first dose of IMP to the first objective tumor progression (progressive disease per RECIST v1.1) or death from any cause, whichever occurs first
Part 1 and Part 2 - Depth of Response | Up to approximately 2 years
  Defined as the maximum percent reduction from baseline in tumor size measured by sum of target lesion diameter (including nodal [short axis] and non-nodal [longest axis] lesions)
Part 1 and Part 2 - Disease Control Rate (DCR) | Up to approximately 2 years
  Defined as the proportion of participants with confirmed CR, confirmed PR, or stable disease (per RECIST v1.1 based on the investigator's assessment) as best overall response
Part 1 and Part 2 - Time to Response (TTR) | Up to approximately 2 years
  Defined as the time from first dose of IMP to first objective response (CR or PR per RECIST v1.1 based on the investigator's assessment)
Part 1 and Part 2 - Overall Survival (OS) | Up to approximately 2 years
  Defined as the time from first dose of IMP to death from any cause
Part 1 and Part 2 - PK assessment: Maximum concentration (Cmax) derived from serum concentration of pumitamig | from pre-dose to the end of study treatment (up to approximately 2 years)
Part 1 and Part 2 - Number of participants developing detectable anti-pumitamig antibodies in serum | from pre-dose to the end of study treatment (up to approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (23):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - NYU Langone - NYU Grossman School of Medicine, New York, New York
  - Texas Oncology, P.A., Houston, Texas
- Australia (2):
  - Cancer Research SA (CRSA), Adelaide, South Austraila
  - One Clinical Research - Hollywood Private Hospital, Nedlands, Western Australia
- South Korea (4):
  - Gyeongsang National University Hospital (GNUH), Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- Turkey (Türkiye) (5):
  - Baskent University Adana Turgut Noyan Application and Research Center Kisla Health Campus, Adana
  - Memorial Ankara Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Memorial Antalya Hospital, Antalya
  - Yeditepe University Hospital, Istanbul
- United Kingdom (4):
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff
  - St James's University Hospital - Leeds Teaching Hospitals NHS Trust, Leeds
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No